CLINICAL TRIAL: NCT00620919
Title: RG1068 (Synthetic Human Secretin) Enhanced Multidetector CT Pancreatography: Evaluation of the Pancreatic Duct in Patients With Known or Suspected Chronic Pancreatitis
Brief Title: Secretin Enhanced Multidetector CT Pancreatography for Evaluation of Known or Suspected Chronic Pancreatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor patient enrollment due to logistical issues.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Dr. Dushyant Sahani, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006P002501
Record Dates: First submitted 2008-01-22; First posted 2008-02-22 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Drug + MDCT
  Interventions: Drug: RG1068 (Synthetic Human Secretin)

INTERVENTIONS:
Drug: RG1068 (Synthetic Human Secretin) — Dose: 0.2 μg/kg of synthetic human or 18.5 µg for patients over 50 kg Route: Intravenous Frequency: Once Duration: Over 1 minute

SUMMARY:
1. To assess the effect of RG1068 at a dose of 0.2 mcg/kg intravenously (IV) on the diameter of the pancreatic duct when used during Multidetector Computed Tomography (MDCT) of the pancreas.
2. To demonstrate that RG1068-enhanced MDCT improves image quality of the pancreas in patients with chronic pancreatitis.
3. To evaluate if RG1068 enhanced MDCT results in improved delineation of structural abnormalities of the pancreatic duct as compared to non-enhanced MDCT.

DETAILED DESCRIPTION:
Multidetector Computed Tomography (MDCT) is the mainstay of imaging for patients with acute or chronic pancreatitis, suspected pancreatic neoplasms and post-pancreatic surgery evaluation. The use of multidetector row helical CT scanners and sub-second gantry rotations, have dramatically reduced scan acquisition time with resultant improvement in patient compliance and image quality. The improved Z-axis (isotropic) resolution permits excellent image reconstructions, which play a critical role in diagnosis and staging of pancreatic pathologies, due to the anatomic layout of the pancreas and its vasculature. Fast scanning time enables the acquisition of multiple phases of enhancement, which is of paramount importance in imaging the pancreas [1].

Until relatively recently, endoscopic retrograde cholangiopancreatography (ERCP) was the primary diagnostic and therapeutic modality for assessing patients with suspected pancreatic disease or abnormalities. However, this invasive procedure carries with it a significant potential for complications including acute pancreatitis, hemorrhage and infection, as well as reactions to contrast material or premedications and exposure to radiation. In addition, the success of such procedures - both from the standpoint of safety and efficacy - is highly dependent on the skill of the endoscopist [2], and the cost of ERCP is relatively high.

Secretin enhanced MRCP (S-MRCP) has been extensively used in assessment of suspected pancreatic diseases. Likewise, administration of secretin intravenously to patients undergoing MDCT for the pancreas will result in improved distension of the pancreatic duct. The potential benefits of this would be a non-invasive evaluation of the pancreatic duct morphology. In patients with suspected abnormality involving the main duct or its side branches, the improved distension of the duct is likely to improve diagnostic yield for conditions such as intraductal papillary mucinous neoplasms (IPMNs) and cystic pancreatic neoplasms.

This study is being undertaken to prospectively assess the effectiveness of RG1068-enhanced MDCT relative to unenhanced MDCT. RG1068 is a synthetic human secretin with a pharmacological profile very similar to that of biological and synthetic porcine secretins. Secretin is a 27-amino acid gastrointestinal peptide hormone that is produced by S-cells in the duodenum in response to the pH decrease caused by the passage of partially digested food from the stomach into the intestine. RG1068 is identical in amino acid sequence to naturally occurring human secretin and differs from porcine secretin in 2 amino acids.

ELIGIBILITY:
Inclusion Criteria:

* Males and females older than 18 years of age
* Is clinically indicated for contrast-enhanced MDCT of the pancreas
* Scheduled for MDCT and therapeutic or diagnostic ERCP for the assessment of chronic pancreatitis
* Has been fully informed and has personally signed and dated the Written Informed Consent and Health Insurance Portability Accountability Act (HIPAA) provisions
* Is a male, or is a female not of childbearing potential, or is a female of childbearing potential who is using effective contraception and has a negative urine pregnancy test on the same day, but prior to, study drug administration
* Is able and willing to complete all study procedures specified in the protocol

Exclusion Criteria:

* Has no clear written indication for contrast enhanced MDCT of the pancreas
* Has a history of hypersensitivity to iodine-containing compounds
* Has congestive cardiac failure (class III-IV in accordance with the classification of the New York Heart Association [NYHA])
* Presence of a pancreatic stent
* Is unable to comply with the study requirements including follow-up
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease which, in the opinion of the investigator, precludes study participation
* History of sensitivity to any of the ingredients in the study drug
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
MDCT-Images will be evaluated for quality, main and branch duct visualization, ductal diameter and improved visualization of structural abnormalities with and without use of RG1068. | 1

SECONDARY OUTCOMES:
Laboratory | 2

CONTACTS AND LOCATIONS:
Overall Officials: Dushyant V Sahani, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States